CLINICAL TRIAL: NCT03277040
Title: DEAL Trial: Diet, Eating, and Lifestyle Improvement for Valued Employees and Their Relatives
Brief Title: Diet, Eating, and Lifestyle Improvement for Valued Employees and Their Relatives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Carolyn Cannuscio, Assistant Professor of Family Medicine and Community Health, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 827780
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Diet Habit; Obesity; Food Habits
MeSH Terms: conditions — Feeding Behavior; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (CSA membership) (Experimental): Employees will gain CSA membership - they will receive bi-weekly deliveries of fresh fruits and vegetables to a central location near their place of employment.
  Interventions: Other: CSA membership
- Control (no CSA membership) (No Intervention): Usual care, usual employee benefits. Employees do not gain CSA membership.

INTERVENTIONS:
Other: CSA membership — Bi-weekly fresh food delivery
  Arms: Intervention (CSA membership)

SUMMARY:
Food is widely understood as a cornerstone of health, however multiple barriers stand between well-intentioned, well-informed consumers and the adoption of healthier dietary practices. This mixed-methods randomized controlled trial (RCT) will measure the impact of offering a Community Sustained Agriculture (CSA) share as an employee benefit on household food environments (diets), eating behaviors, and lifestyles.

DETAILED DESCRIPTION:
Aim: We will test a strategy to increase frequency of cooking meals at home and consumption of healthful, fresh foods by providing study participants with a CSA membership.

Study design: This is a mixed method randomized controlled trial, with survey, home-food audit, and interview components.

Hypothesis: The intervention group who received a CSA membership as an employee benefit will prepare more meals at home and consume more healthful, fresh foods compared to the control group (no CSA participation).

Using both qualitative and quantitative assessments, outcomes will be measured using 3 primary measures:

1. Home food audits at baseline and at week 8 of the intervention. A random selection of participants will have home-food audits completed by members of the research team - those not randomly selected will complete the home-food audit themselves.
2. Self-administered surveys, including food frequency questionnaires, at baseline, week 8, and week 16.
3. Randomly selected participants will be asked to participate in qualitative interviews at the close of the 16-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are non-faculty employees at the University of Pennsylvania and University of Pennsylvania Health System.
* Individuals who score below the median (50th percentile) on dinners prepared at home on screening survey.

Exclusion Criteria:

* Individuals who are under the age of 18.
* Individuals who are already have a CSA membership.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Quantity of meals prepared and consumed at home. | 16 Weeks

SECONDARY OUTCOMES:
Self-reported satisfaction with employee benefits | 16 Weeks
Time spent planning meals | 16 Weeks
Time spent preparing meals | 16 Weeks
Perceived stress regarding food shopping, meal planning, and meal preparation | 16 Weeks
  Perceived stress regarding food shopping, meal planning, and meal preparation, assessed during follow-up qualitative interviews
Perceived stress regarding food shopping, meal planning, and meal preparation | 16 Weeks
  Perceived stress regarding food shopping, meal planning, and meal preparation, measured comparing baseline and follow-up surveys using likert scale questions
Knowledge and self-efficacy regarding healthy food preparation | 16 Weeks
  Knowledge and self-efficacy regarding healthy food preparation, assessed during follow-up qualitative interviews
Knowledge and self-efficacy regarding healthy food preparation | 16 Weeks
  Knowledge and self-efficacy regarding healthy food preparation, measured comparing baseline and follow-up surveys using likert scale questions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feuerstein-Simon R, Dupuis R, Schumacher R, Cannuscio CC. A Randomized Trial to Encourage Healthy Eating Through Workplace Delivery of Fresh Food. Am J Health Promot. 2020 Mar;34(3):269-276. doi: 10.1177/0890117119890804. Epub 2019 Dec 16. PMID 31840522